CLINICAL TRIAL: NCT05543629
Title: A Phase 1b/2 Study of BMS-986442 in Combination With Nivolumab or Nivolumab and Chemotherapies in Participants With Advanced Solid Tumors and Non-small Cell Lung Cancer
Brief Title: A Study of BMS-986442 With Nivolumab With or Without Chemotherapy in Solid Tumors and Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA115-001; 2022-501676-26 (EudraCT Number); U1111-1283-1243 (Registry Identifier: WHO)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors; Non-small Cell Lung Cancer
Keywords: BMS-986442; Nivolumab; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Docetaxel; taxane; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: BMS-986442 + Nivolumab (Experimental)
  Interventions: Biological: BMS-986442; Biological: Nivolumab
- Part B1: BMS-986442 + Nivolumab (Experimental): Second line (2L) + Post-immuno-oncology (IO)/Platinum-Doublet Non-small cell lung cancer (NSCLC)
  Interventions: Biological: BMS-986442; Biological: Nivolumab
- Part B2: BMS-986442 + Nivolumab (Experimental): Post IO Gastric Cancer/Gastroesophageal Junction and Post-IO squamous cell carcinoma of the head and neck (SCCHN)
  Interventions: Biological: BMS-986442; Biological: Nivolumab
- Part C: BMS-986442 + Nivolumab + Docetaxel (Experimental)
  Interventions: Biological: BMS-986442; Biological: Nivolumab; Drug: Docetaxel
- Part D: BMS-986442 + Nivolumab + Carboplatin + Pemetrexed (Experimental)
  Interventions: Biological: BMS-986442; Biological: Nivolumab; Drug: Carboplatin; Drug: Pemexetred
- Part E: BMS-986442 + Nivolumab + Carboplatin + Paclitaxel (Experimental)
  Interventions: Biological: BMS-986442; Biological: Nivolumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: BMS-986442 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Drug: Docetaxel — Specified dose on specified days
  Other Names: Taxane / Toxotere chemotherapy
  Arms: Part C: BMS-986442 + Nivolumab + Docetaxel
Drug: Carboplatin — Specified dose on specified days
  Other Names: Platinum chemotherapy
  Arms: Part D: BMS-986442 + Nivolumab + Carboplatin + Pemetrexed; Part E: BMS-986442 + Nivolumab + Carboplatin + Paclitaxel
Drug: Pemexetred — Specified dose on specified days
  Other Names: Folate analog metabolic inhibitor
  Arms: Part D: BMS-986442 + Nivolumab + Carboplatin + Pemetrexed
Drug: Paclitaxel — Specified dose on specified days
  Other Names: Taxane chemotherapy
  Arms: Part E: BMS-986442 + Nivolumab + Carboplatin + Paclitaxel

SUMMARY:
The purpose of this study is to evaluate BMS-986442 in combination with nivolumab (with or without chemotherapy) for its antitumor efficacy and benefit to participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants in all parts of the study must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participants must have a life expectancy of at least 3 months at the time of first dose.

Exclusion Criteria:

* Untreated symptomatic central nervous system metastases or leptomeningeal metastases.
* Concurrent malignancy (present during screening) requiring treatment, or history of prior malignancy active within 2 years prior to randomization in study Part B1 or treatment assignment in all other study parts.
* Participants with an active, known, or suspected autoimmune disease.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (14):
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - Local Institution - 0096, Costa Mesa, California
  - Local Institution - 0075, Orange, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Local Institution - 0027, Orlando, Florida
  - Local Institution - 0029, Fort Wayne, Indiana
  - Local Institution - 0022, New Orleans, Louisiana
  - Local Institution - 0005, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Local Institution - 0003, Hackensack, New Jersey
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Local Institution - 0019, Cincinnati, Ohio
  - Local Institution - 0046, Allentown, Pennsylvania
  - Local Institution - 0016, Houston, Texas
- Australia (5):
  - Local Institution - 0018, Darlinghurst, New South Wales
  - Local Institution - 0001, Westmead, New South Wales
  - Local Institution - 0086, Southport, Queensland
  - Local Institution - 0002, Clayton, Victoria
  - Local Institution - 0084, Murdoch, Western Australia
- Italy (4):
  - Local Institution - 0065, Milan, Milano
  - Local Institution - 0064, Candiolo, Torino
  - Local Institution - 0077, Siena, Tuscany
  - Local Institution - 0062, Napoli
- Poland (3):
  - Local Institution - 0067, Warsaw, Masovian Voivodeship
  - Local Institution - 0073, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0069, Bydgoszcz
- Spain (6):
  - Local Institution - 0080, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0083, Madrid, Madrid, Comunidad de
  - Local Institution - 0079, Madrid, Madrid, Comunidad de
  - Local Institution - 0082, Málaga
  - Local Institution - 0087, Seville
  - Local Institution - 0081, Valencia

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Treatment 1: BMS-986442 20mg + Nivo 360mg QW
- Part A: Treatment 2: BMS-986442 60mg + Nivo 360mg QW
- Part A: Treatment 3: BMS-986442 200mg + Nivo 360mg QW
- Part A: Treatment 4; Part B1: Treatment 1: BMS-986442 600mg + Nivo 360mg QW
- Part A: Treatment 5; Part B1: Treatment 2; Part B2: Treatment 1: BMS-986442 1200mg + Nivo 360mg QW
Period: Overall Study
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Started | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by Sponsor | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Not completed — Not Reported | 2 | 2 | 0 | 0 | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1 | Total
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (7.50) | 66.3 (1.15) | 66.2 (7.41) | 76.3 (3.79) | 57.3 (9.71) | 65.3 (8.86) | 60.1 (11.41) | 65.7 (1.53) | 63.7 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 3 | 1 | 5 | 0 | 18
  Male | 2 | 2 | 1 | 1 | 0 | 6 | 3 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 4 | 3 | 3 | 7 | 8 | 2 | 34
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  White | 4 | 3 | 3 | 2 | 1 | 7 | 7 | 2 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events.
  An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
  An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
  For the reporting of all AEs, including intensity or severity, on case report forms, please follow the definitions in National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (NCI CTCAE v5).
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Participants | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death.
  * Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Participants | 3 | 0 | 4 | 2 | 1 | 4 | 6 | 1

3. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: Number of Participants with adverse events leading to discontinuation
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: DLTs will be defined based on the incidence, intensity, and duration of the AEs for which no clear alternative cause is identified and will exclude events clearly related to disease progression or intercurrent illness.
  in addition, the following AEs will be DLTs:
  * Any death that is not clearly due to the underlying disease or extraneous causes
  * Any Grade ≥ 3 non-hematological toxicity
  * Any Grade myocarditis
  * Any Grade myelitis, encephalitis, myasthenia gravis, or Guillain-Barre syndrome
  * Grade 4 neutropenia of > 7 days duration
  * Grade 4 thrombocytopenia.
  * Grade 3 thrombocytopenia with clinically significant bleeding.
  * Febrile neutropenia
  Any AE that is not clearly due to disease progression or extraneous causes that occurs within the 28-day DLT evaluation window and meets criteria for permanent discontinuation will be considered a DLT.
Time Frame: From Cycle 1 day 1 to day 28 (28 Days)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants Who Died
Description: Number of Participants who died
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Participants | 2 | 0 | 3 | 0 | 1 | 1 | 2 | 2

6. Secondary Outcome: CMax
Description: Maximum observed serum concentration
Time Frame: On Cycle 1 Day 1 and on Cycle 4 Day 1 (Each cycle = 3 Weeks)
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 6 | 3
  Cycle 1 Day 1 | 6.47 (12.07) | 20.66 (31.27) | 84.64 (12.90) | 213.29 (24.73) | 607.16 (30.57) | 188.17 (12.48) | 525.77 (63.12) | 278.89 (9.14)
  Cycle 4 Day 1: number analyzed (Participants) | 3 | 1 | 2 | 1 | 1 | 2 | 3 | 0
  Cycle 4 Day 1 | 7.53 (13.81) | 28.60 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 88.92 (26.63) | 239.00 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 595.00 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 161.37 (20.29) | 345.40 (25.64) |

7. Secondary Outcome: Tmax
Description: Time of maximum observed serum concentration
Time Frame: On Cycle 1 Day 1 and on Cycle 4 Day 1 (Each cycle = 3 Weeks)
Population: PK evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
hours
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 6 | 3
  Cycle 1 Day 1 | 4.0 [1.0 to 4.0] | 1.17 [1.0 to 2.7] | 1.52 [1.2 to 2.5] | 1.77 [1.0 to 2.1] | 4.05 [0.3 to 22.4] | 1.27 [1.0 to 4.0] | 1.67 [1.0 to 4.0] | 1.67 [1.5 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 3 | 1 | 2 | 1 | 1 | 2 | 3 | 0
  Cycle 4 Day 1 | 1.22 [1.0 to 3.0] | 3.88 [3.88 to 3.88] | 1.23 [1.1 to 1.4] | 3.93 [3.93 to 3.93] | 23.98 [23.98 to 23.98] | 13.94 [3.0 to 24.9] | 5.50 [3.9 to 5.5] |

8. Secondary Outcome: AUC (Tau)
Description: Area under the serum concentration-time curve in 1 dosing interval
Time Frame: On Cycle 1 Day 1 and on Cycle 4 Day 1 (Each cycle = 3 Weeks)
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
h*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 6 | 3
  Cycle 1 Day 1 | 697.89 (22.59) | 2182.10 (60.66) | 10412.98 (19.48) | 31421.18 (14.61) | 92086.95 (42.72) | 23544.68 (21.49) | 59747.91 (26.15) | 28983.46 (22.78)
  Cycle 4 Day 1: number analyzed (Participants) | 3 | 1 | 2 | 1 | 1 | 1 | 3 | 0
  Cycle 4 Day 1 | 650.12 (91.31) | 4048.56 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 6965.42 (24.78) | 42581.54 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 129835.00 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 31371.02 (NA) — Insufficient number of participants analyzed to calculate geometric coefficient of variation | 42688.89 (19.18) |

9. Secondary Outcome: Number of Participants With BMS-986442 Anti Drug Antibody (ADA)
Description: Number of participants with BMS-986442 Anti Drug Antibody (ADA)
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants with baseline and at least one post-baseline evaluable ADA assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 2 | 7 | 7 | 2
Participants
  Baseline ADA Positive: number analyzed (Participants) | 5 | 3 | 4 | 3 | 2 | 7 | 6 | 2
  Baseline ADA Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Positive | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
  ADA Persistent Positive | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  ADA Not PP- Last sample postive | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Other Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Negative | 5 | 2 | 3 | 3 | 1 | 6 | 5 | 2

10. Secondary Outcome: Objective Response Rate (ORR) Per Recist v1.1 by Investigator
Description: ORR is defined as the number of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) assessed by Investigator, according to RECIST v1.1 criteria, divided by the number of treated participants.
  The BOR is defined as the best response designation recorded between the date of first dose and the date of initial objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. For purposes of analysis, if a participant receives one dose and discontinues the study without assessment or receives subsequent therapy prior to assessment, this participant will be counted in the denominator (as nonrespondent).
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Percentage of Participants | 20.0 [0.5 to 71.6] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9] | 0 [0.0 to 70.8]

11. Secondary Outcome: Disease Control Rate (DCR) Per Recist v1.1 by Investigator
Description: Disease Control Rate (DCR) is defined as the number of treated participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD) (and/or SD > 6 months), based on investigator assessments divided by the number of all treated participants.
Time Frame: From first dose to 100 days post last dose (Approximately 6 Months)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 3 | 7 | 8 | 3
Percentage of Participants | 20.0 [0.5 to 71.6] | 0 [0.0 to 70.8] | 25.0 [0.6 to 80.6] | 0 [0.0 to 70.8] | 66.7 [9.4 to 99.2] | 14.3 [0.4 to 57.9] | 12.5 [0.3 to 52.7] | 33.3 [0.8 to 90.6]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately on average up to 6 months with a maximum of 16 months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Part A: Treamtent 5; Part B1: Treatment 2; Part B2: Treatment 1: BMS-986442 1200mg + Nivo 360mg QW
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treamtent 5 | Part B1: Treatment 1 | Part B1: Treatment 2 | Part B2: Treatment 1
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/3 | 3/4 | 0/3 | 1/3 | 1/7 | 2/8 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/5 | 0/3 | 4/4 | 2/3 | 1/3 | 4/7 | 6/8 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 4/4 | 3/3 | 3/3 | 7/7 | 7/8 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment 1 (N=5) | Part A: Treatment 2 (N=3) | Part A: Treatment 3 (N=4) | Part A: Treatment 4 (N=3) | Part A: Treamtent 5 (N=3) | Part B1: Treatment 1 (N=7) | Part B1: Treatment 2 (N=8) | Part B2: Treatment 1 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0 | 0 | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment 1 (N=5) | Part A: Treatment 2 (N=3) | Part A: Treatment 3 (N=4) | Part A: Treatment 4 (N=3) | Part A: Treamtent 5 (N=3) | Part B1: Treatment 1 (N=7) | Part B1: Treatment 2 (N=8) | Part B2: Treatment 1 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 4 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perineal rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 2 | 2 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT05543629/Prot_SAP_000.pdf